CLINICAL TRIAL: NCT04937543
Title: Randomized, Open-label, Three Arms Study to Evaluate the Efficacy of Inhaled Therapies in the Treatment of Acute Symptoms Associated With COVID-19 and in the Prevention of the Use of Health Resources in Patients With ≥ 18 Years Old (TRIVID Study)
Brief Title: Efficacy of Inhaled Therapies in the Treatment of Acute Symptoms Associated With COVID-19
Acronym: TRIVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIV001
Record Dates: First submitted 2021-06-23; First posted 2021-06-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Covid19
Keywords: SARS-CoV-2; corticosteroids; Bronchodilators
MeSH Terms: conditions — COVID-19 | interventions — Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No intervation (No Intervention): patients receiving standart of care
- Experimental intervation one (Active Comparator): patients receiving standart of care + inhaled beclometasone
  Interventions: Drug: inhaled beclametasone
- Experimental intervation two (Active Comparator): patients receiving standart of care + inhaled beclometasone/ formoterol / glycopyrronium
  Interventions: Drug: Inahaled beclomethasone / formoterol / glycopyrronium

INTERVENTIONS:
Drug: inhaled beclametasone — Adding belcamethasone to standard of care for Covid 19 positive patients
  Arms: Experimental intervation one
Drug: Inahaled beclomethasone / formoterol / glycopyrronium — Adding belcametasone/ formoterol / glycopyrronium to standard of care for Covid 19 positive patients
  Arms: Experimental intervation two

SUMMARY:
Introduction: SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2), the new coronavirus, causes a disease called COVID-19 that can trigger aggressive inflammatory responses. In this sense, inhaled corticosteroid therapy (IC) has shown some favorable results in controlling the worsening of the disease, given that it has effects on pulmonary inflammation and can be an intervention to be used in the mild manifestations of COVID-19 in order to prevent disease progression and severity. Regarding the role of bronchodilators, studies have suggested that their combination with IC exerts synergistic therapeutic effects. Objective: To determine the efficacy of inhaled therapy of beclomethasone/formoterol/glycopyrronium (BFG) (100/6/12.5mcg) and/or beclomethasone HFA 250 mcg in preventing the use of healthcare resources in patients ≥ 18 years of age at 28 days compared to usual care. Method: participants will be randomized according to a ratio of 1:1:1 into three groups: (Group 1) Standard of care + BFG two doses 2x/day; (Group 2) standard treatment + beclomethasone HFA two doses 2x/day and (Group 3) standard treatment. After collecting the signed informed consent form, research participants will be treated for 28 days and, after two days, will undergo a spirometry test. Therefore, the total duration of the study for a given participant will be up to 30 days.

ELIGIBILITY:
Inclusion Criteria: A research participant will be eligible to participate in this study if ALL of the following criteria are met:

1. Adult men or women (≥ 18 years of age)
2. PCR positive SarsCoV-2
3. Symptomatic participants must have at least 1 of the following symptoms in the inclusion: fever or self-reported fever perception in the last 24 hours, headache, sore throat, dry cough, fatigue, chest pain or choking sensation (without associating to respiratory distress), myalgia, anosmia, ageusia or gastrointestinal symptoms with up to 10 days onset.
4. Participants with arterial pulse oximetry (SpO2) saturation ≥ 92% in room air at inclusion.
5. Participants with the following hematological and biochemical laboratory parameters obtained in the period of 7 days before D0:

   * Hemoglobin> 9.0 g / dL-1
   * Absolute Neutrophil Count ≥ 1000 mm-³
   * Platelets ≥ 100,000 mm-3
   * Creatinine clearance ≥ 30 mL / min-1 using the Cockcroft-Gault formula
   * Alkaline phosphatase <10 × upper limit of normal (LSN), AST (TGOS) and ALT (TGPS) <10 × LSN.
   * Laboratory pregnancy test (Negative β-hCG).
6. Participants must understand, sign and date the voluntary informed consent form in writing at the visit prior to any specific protocol procedure.
7. Participants must be able and willing to comply with study visits and procedures, as per the protocol.

Exclusion Criteria:

Research participants who meet any of the following exclusion criteria will be excluded from the study:

1. Participants with moderate or severe acute respiratory failure or needing non-invasive ventilation or oxygen, or with SpO2 <92% or tachypnea (respiratory rate ≥ 30 breaths / minute).
2. Participants with pre-existing, severe and uncontrolled organ failure, which prevents participation in the study by the investigator's judgment (non-relevant cardiac disease)
3. Participant diagnosed with previous asthma using inhaled or oral corticosteroids in the last four weeks.
4. Participant with previous use, in the last ten days of randomization, of inhaled, oral or injectable corticosteroids.
5. Participant with previous diagnosis of chronic obstructive pulmonary disease, even if he is not using any inhaled medication.
6. Pregnant or lactating women.
7. Use of any product under investigation or unregistered within 3 months or within 5 half-lives before baseline, whichever is longer.
8. Hypersensitivity to the drug and / or its excipients.
9. Any condition that, in the investigator's opinion, could compromise the participant's safety or his adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in preventing the use of health resources in patients | 28 days after treatment

SECONDARY OUTCOMES:
Airway obstruction | 28 days after treatment
  Spirometry
Small airway obstruction | 28 days after treatment
  computadorized tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided